CLINICAL TRIAL: NCT02656095
Title: Lipoprotein Lipase Enzyme Activity Assay Validation and Clinical Assessment
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1412; UL1TR001082 (NIH)
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Lipoprotein Lipase Deficiency
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Heparin — Participants will be given IV heparin in order to release lipoprotein lipase from capillary endothelial cells. Blood will be drawn 10-15 minutes post-heparin administration and run through assay to determine lipoprotein lipase levels.

SUMMARY:
This study plans to learn more about measuring Lipoprotein lipase (LPL) activity in humans. LPL is an enzyme in the breakdown of certain types of fats into smaller parts. Lipoprotein lipase deficiency (LPLD) is a very rare genetic disorder in which lipoprotein enzyme is no longer functional. This can cause conditions known as high triglycerides in the blood and inflammation of the pancreas.

Investigational medications to treat LPLD are currently being developed. In order to see if these medications are effective, it is necessary to be able to accurately measure LPL activity in humans.

LPL activity has been successfully measured in animal models after giving heparin. Heparin is a blood thinner which is approved by the FDA. It is originally used to prevent blood clots. This study will administer heparin to healthy adults through intravenous infusion (IV). Blood samples will be collected before and after the infusion to test LDL levels.

The purpose of this study is to develop a cheap, more reliable standard for assessment of LPLD in patients

ELIGIBILITY:
Inclusion Criteria:

1. male and females between ages of 20-39

Exclusion Criteria:

1. Past history of LPL deficiency
2. Hypercholesterolemia (Cholesterol >200, LDL >160, HDL <35) hypertriglyceridemia (TG>150), any familial lipid disorder
3. Diabetes mellitus (type 1 or 2)
4. Uncontrolled hypertension SBP>140, DBP>90
5. History of hemorrhagic stroke
6. Current pregnancy
7. History of major surgery, invasive procedure or trauma within the last 30 days, or planned major surgery within 30 days after participating in the study
8. Exposure to heparin (unfractionated heparin or low molecular weight heparin) within 30 days prior to screening
9. History of allergy to heparin
10. History of heparin-induced thrombocytopenia
11. Current smoking
12. Active ulcerative or angiodysplastic GI diseases
13. Thrombocytopenia or platelet disorders (Platelet count <100,000/UL)
14. Major health issues which may affect the safety of study subject, including but not limited to:

    * History of chronic kidney disease (eGFR<60)
    * Long term use of medications which alter lipid metabolism
    * History of hepatic disease (ALT or AST more than 2 times the upper limit of normal)
    * History of clotting disorders, any type of coagulation factor deficiency, or thrombocytopenia
    * Chronic use of ASA, anticoagulants, platelet inhibitors
    * Use of NSAIDS for more than 2 weeks prior to screening
    * Anemia (hemoglobin <13 g/dL)

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Male and female individuals
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Lipoprotein lipase levels | 10-15 minutes post-heparin adminstration
  Blood will be drawn after IV heparin administration and run through assay to determine lipoprotein lipase levels.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Eckel, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No